CLINICAL TRIAL: NCT00433654
Title: EnRhythm MRI™ SureScan™ Pacing System Clinical Investigation
Brief Title: EMRI SureScan™ Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 212
Record Dates: First submitted 2007-02-02; First posted 2007-02-12 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2011-07

CONDITIONS: Bradycardia; Slow Heart Beat
Keywords: Bradycardia; Slow heart beat; Magnetic resonance imaging (MRI)
MeSH Terms: conditions — Bradycardia | interventions — Bone Wires; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI group (Active Comparator): The MRI group underwent a one-hour MRI scan at the 9-12 weeks post-implant follow-up.
  Interventions: Device: Implantable Pulse Generator (IPG) and Pacing Leads (wires); Other: Magnetic Resonance Imaging (MRI) scan
- Control group (Other): The control group waited for one hour (no MRI) at the 9-12 weeks post-implant follow-up.
  Interventions: Device: Implantable Pulse Generator (IPG) and Pacing Leads (wires)

INTERVENTIONS:
Device: Implantable Pulse Generator (IPG) and Pacing Leads (wires) — Pacer and leads
Other: Magnetic Resonance Imaging (MRI) scan — One hour MRI scan on the head and lower back.
  Arms: MRI group

SUMMARY:
The purpose of this clinical study is to confirm safety and efficacy in the clinical magnetic resonance imaging (MRI) environment of the investigational EnRhythm MRI™ SureScan™ Pacing System (used in support of Revo MRI™ SureScan Pacing System launch).

DETAILED DESCRIPTION:
This study is a prospective, multi-center global study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has, or is at risk of having, a heart beat that is too slow and his/her doctor has determined he/she needs a pacemaker.
* Subject available for follow-up at study center for length of study.
* Subject able and willing to undergo elective MRI scanning without sedation.

Exclusion Criteria:

* Subject has, or is at risk of having, a heart beat that is too fast and his/her doctor has determined he/she needs an implantable cardioverter defibrillator (ICD).
* Subject needs or will need another MRI-scan, other than those required by the study, during the required study follow-up period.
* Pregnant women, or women of child bearing potential who are not on a reliable form of birth control.
* Subject with exclusion criteria required by local law.
* Subject who intends to participate in another clinical study during this clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: EMRI SureScan Clinical Study Team, Study Chair — Medtronic
Locations (45):
- United States (15):
  - Redwood City, California
  - Salinas, California
  - Orlando, Florida
  - Peachtree City, Georgia
  - Des Moines, Iowa
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Mineola, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Erie, Pennsylvania
  - Knoxville, Tennessee
  - Charlottesville, Virginia
  - Norfolk, Virginia
- Austria (2):
  - Graz
  - Linz
- Belgium (2):
  - Liège
  - Mons
- Canada (6):
  - Calgary, Alberta
  - Victoria, British Columbia
  - Kingston, Ontario
  - London, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
- Prague, Czechia
- Rouen, France
- Germany (10):
  - Bad Nauheim
  - Bonn
  - Dortmund
  - Dresden
  - Essen
  - Göttingen
  - Hamburg
  - Marburg
  - München
  - Ulm
- Italy (4):
  - Asti
  - Pescia
  - Pietra Ligure
  - Viterbo
- Netherlands (2):
  - Amsterdam
  - Nieuwegein
- Zurich, Switzerland
- London, United Kingdom

REFERENCES:
- [Derived] Sutton R, Kanal E, Wilkoff BL, Bello D, Luechinger R, Jenniskens I, Hull M, Sommer T. Safety of magnetic resonance imaging of patients with a new Medtronic EnRhythm MRI SureScan pacing system: clinical study design. Trials. 2008 Dec 2;9:68. doi: 10.1186/1745-6215-9-68. PMID 19055703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first implant occurred 5 February 2007. A total of 484 subjects were enrolled, including 113 enrollments at 13 centers in the US and 371 enrollments at 29 centers outside of the US.
Pre-assignment Details: Implant procedure included EnRhythm MRI SureScan pacemaker and 2 CapsureFix MRI 5086MRI leads. Pacemaker function and adverse events were assessed. 17 subjects did not have an implant attempt. 3 subjects received a subset of the 3 system components and were followed for safety. All other subjects were randomized after successful implant.
Groups:
- MRI Group: The MRI group underwent a one-hour MRI scan at 9-12 weeks post-implant.
- Control Group: The control group waited for one hour (no MRI scan) at 9-12 weeks post-implant
Period: Overall Study
Arm/Group | MRI Group | Control Group
Started | 258 | 206
Completed | 243 (Subjects completing the 4-month follow-up.) | 201 (Subjects completing the 4-month follow-up.)
Not Completed | 15 | 5
Not completed — Death | 4 | 0
Not completed — Missed visit | 6 | 3
Not completed — Subject not yet due for visit | 4 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Control Group: The control group waited for one hour (did not have an MRI scan) at 9-12 weeks post-implant.
- Total: Total of all reporting groups
Arm/Group | MRI Group | Control Group | Total
Number analyzed (Participants) | 258 | 206 | 464
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 67 | 142
  >=65 years | 183 | 139 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (12.9) | 68.0 (12.6) | 68.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 71 | 175
  Male | 154 | 135 | 289
Region of Enrollment [Number; unit: participants]
  United States | 66 | 33 | 99
  Europe | 157 | 141 | 298
  Canada | 34 | 32 | 66
  Middle East | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Magnetic Resonance Imaging (MRI)-Related Complications
Description: Subjects with a complication related to the MRI scan. All adverse events in the time frame were recorded at the subject's center and assessed by a centralized Adverse Event Advisory Committee. The committee determined whether each adverse event was a complication (requiring invasive intervention), and whether the event was related to the MRI scan.
Time Frame: MRI scan to one-month post-MRI scan
Population: Subjects who underwent an MRI scan following study protocol-specified instructions are included. Of the 243 subjects who completed a one-month post-MRI (4-month) visit, 32 did not complete the MRI scan according to the protocol instructions, and are not included.
Measure: Number; unit: participants
Arm/Group | MRI Group
Number analyzed (Participants) | 211
participants | 0
Statistical Analysis 1: Comparison: MRI Group; Null hypothesis: rate > 10%; Test type: Superiority or Other; p < 0.001, exact test of binomial proportions; Percentage = 0, 95% CI 1-sided [upper limit 1.7]

2. Primary Outcome: Atrial Pacing Capture Threshold Success
Description: Subjects' atrial pacing capture threshold (the energy sent from the pacemaker needed to make the heart's atrium beat) was measured at the 9-12 week visit (before the MRI scan was performed for those in the MRI group) and at the 4-month visit (one month post-MRI). Subjects were considered successful if their pacing capture threshold did not increase by 1.0 volt (V) or more.
Time Frame: 9-12 week visit to 4-month visit
Population: Subjects were excluded from this analysis if: they did not have atrial pacing capture threshold measurements at 9-12 weeks or 4 months; or (for the MRI group) their MRI scan was not done according to protocol.
Measure: Number; unit: participants
Groups:
- Control Group: The control group waited for one hour (no MRI) at the 9-12 week follow-up.
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 165 | 164
participants | 165 | 164
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: success rate MRI group <= success rate control group - 10%; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 10%; Farrington-Manning — P-value and confidence interval could not be calculated because both groups were 100% successful; Difference in percentages = 0

3. Primary Outcome: Ventricular Pacing Capture Threshold Success
Description: Subjects' ventricular pacing capture threshold (the energy sent from the pacemaker needed to make the heart's ventricle beat) was measured at the 9-12 week visit (before the MRI scan was performed for those in the MRI group) and at the 4-month visit (one month post-MRI). Subjects were considered successful if their pacing capture threshold did not increase by 1.0 volt (V) or more.
Time Frame: 9-12 week visit to 4-month visit
Population: Subjects were excluded from this analysis if: they did not have ventricular pacing capture threshold measurements at 9-12 weeks or 4 months; or (for the MRI group) their MRI scan was not done according to protocol.
Measure: Number; unit: participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 190 | 184
participants | 190 | 183
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: success rate MRI group <= success rate control group - 10%; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 10%; p < 0.001, Farrington-Manning; Difference in percentages = 0.5

4. Primary Outcome: Atrial Sensed Amplitude Success
Description: Subjects' atrial sensed amplitude (the minimum energy produced by the heart's atrium that the pacemaker can sense) was measured at the 9-12 week visit (before the MRI scan was performed for those in the MRI group) and at the 4-month visit (one month post-MRI). Subjects were considered successful if their sensed amplitude did not decrease by more than 50% and remained above 1.5 millivolts (mV).
Time Frame: 9-12 week visit to 4-month visit
Population: Subjects were excluded from this analysis if: they did not have atrial sensed amplitude measurements at 9-12 weeks or 4 months; or (for the MRI group) their MRI scan was not done according to protocol; or if their 9-12 week atrial sensed amplitude was less than 1.5 mV.
Measure: Number; unit: participants
Groups:
- Control Group: The control group waited for one hour (no MRI scan) at the 9-12 week follow-up.
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 131 | 139
participants | 124 | 129
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: success rate MRI group <= success rate control group - 10%; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 10%; p < 0.001, Farrington-Manning; Difference in percentages = 1.9

5. Primary Outcome: Ventricular Sensed Amplitude Success
Description: Subjects' ventricular sensed amplitude (the minimum energy produced by the heart's ventricle that the pacemaker can sense) was measured at the 9-12 week visit (before the MRI scan was performed for those in the MRI group) and at the 4-month visit (one month post-MRI). Subjects were considered successful if their sensed amplitude did not decrease by more than 50% and remained above 5.0 millivolts (mV).
Time Frame: 9-12 week visit to 4-month visit
Population: Subjects were excluded from this analysis if: they did not have ventricular sensed amplitude measurements at 9-12 weeks or 4 months; or (for the MRI group) their MRI scan was not done according to protocol; or if their 9-12 week ventricular sensed amplitude was less than 5.0 mV.
Measure: Number; unit: participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 134 | 136
participants | 130 | 129
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: success rate MRI group <= success rate control group - 10%; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 10%; p < 0.001, Farrington-Manning; Difference in percentages = 2.1

6. Secondary Outcome: Subjects With System-related Complications
Description: Subjects with a complication related to the implanted system, which consisted of the pacemaker, leads to the right chambers of the heart (atrium and ventricle), pacemaker software, and programmer. All adverse events in the time frame were recorded at the subject's center and assessed by a centralized Adverse Event Advisory Committee. The committee determined whether each adverse event was a complication (requiring invasive intervention), and whether the event was related to the system.
Time Frame: Implant to 4 Months
Population: All implanted subjects with either a 4-month follow-up or a system-related complication within the first 4 months post-implant are included.
Measure: Number; unit: participants
Groups:
- Implanted Subjects: All subjects undergoing an implant attempt
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 447
participants | 37
Statistical Analysis 1: Comparison: Implanted Subjects; Null hypothesis: Percentage of subjects with complication > 20%; Test type: Superiority or Other; p < 0.001, exact test of binomial proportions; Percentage = 8.3, 95% CI 1-sided [upper limit 10.7]

7. Secondary Outcome: System Related Adverse Device Effects Due to Labeling Instructions
Description: Number of participants with adverse device effects (ADEs) that resulted from insufficiencies or inadequacies in the instructions for use or deployment of the device, or from user error. ADE's were investigator-reported.
Time Frame: Implant through 18 months post-implant
Population: Includes all subjects undergoing an MRI using the instructions in the protocol.
Measure: Number; unit: participants
Arm/Group | MRI Group
Number analyzed (Participants) | 211
participants | 0

8. Secondary Outcome: Occurrence of Arrhythmias
Description: Number of participants with sustained ventricular arrhythmias or asystole episodes that occurred during the MRI scan that were considered attributable to the MRI scan
Time Frame: During the MRI scan
Population: Arrhythmia was defined as heart rate > 150 beats per minute for > 30 seconds. Asystole was defined as standstill 6 seconds in electrical activity of the heart. Episodes were assessed via pulse oximetry monitoring during MRI scans.
Measure: Number; unit: participants
Arm/Group | MRI Group
Number analyzed (Participants) | 211
participants | 0

9. Secondary Outcome: Atrial Lead Impedance Change
Description: Subjects' atrial lead impedance (a measure of electrical resistance) was measured at the 9-12 week visit (before the MRI scan was performed for those in the MRI group) and at the 4-month visit (one month post-MRI). Both measurements were conducted by the pacemaker. The difference between the two is reported.
Time Frame: 9-12 week visit and 4-month visit
Population: Subjects with non-missing data are included
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 201 | 197
ohms | -0.6 (61.8) | 7.3 (50.4)

10. Secondary Outcome: Ventricular Lead Impedance Change
Description: Subjects' ventricular lead impedance (a measure of electrical resistance) was measured at the 9-12 week visit (before the MRI scan was performed for those in the MRI group) and at the 4-month visit (one month post-MRI). Both measurements were conducted by the pacemaker. The difference between the two is reported.
Time Frame: 9-12 week visit and 4-month visit
Population: Subjects with non-missing data are included
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 201 | 196
ohms | -9.0 (48.5) | -5.7 (51.8)

11. Secondary Outcome: Atrial Lead Handling Rating
Description: Physicians' rated atrial lead handling during the implant on a scale of -3 to +3 where: -3 = well below expectations; -2 = moderately below expectations; -1 = slightly below expectations; 0 = met expectations; +1 = slightly above expectations; +2 = moderately above expectations; and +3 = well above expectations.
Time Frame: During implant
Population: All surveys completed are included
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- 5086 MRI Lead: The 5086 MRI lead was used by all subjects in this study
Arm/Group | 5086 MRI Lead
Number analyzed (Participants) | 212
Units on a scale | 0.53 (1.22)

12. Secondary Outcome: Ventricular Lead Handling Rating
Description: Physicians' rated ventricular lead handling during the implant on a scale of -3 to +3 where: -3 = well below expectations; -2 = moderately below expectations; -1 = slightly below expectations; 0 = met expectations; +1 = slightly above expectations; +2 = moderately above expectations; and +3 = well above expectations.
Time Frame: During implant
Population: All surveys completed are included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 5086 MRI Lead
Number analyzed (Participants) | 211
Units on a scale | 0.58 (1.17)

13. Secondary Outcome: Atrial Pacing Capture Threshold
Description: Average atrial pacing capture threshold. Pacing capture threshold is the energy needed to pace the heart.
Time Frame: 3 or 4 months post-implant
Population: Includes all subjects with data.
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 174 | 175
Volts | 0.78 (0.28) | 0.77 (0.66)

14. Secondary Outcome: Ventricular Pacing Capture Threshold
Description: Average ventricular pacing capture threshold. Pacing capture threshold is the energy needed to pace the heart.
Time Frame: 3 or 4 months post-implant
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 197 | 189
Volts | 0.82 (0.30) | 0.90 (0.70)

15. Secondary Outcome: Atrial Sensed Amplitude
Description: Average atrial sensed amplitude.
Time Frame: 3 or 4 months post-implant
Measure: Mean (Standard Deviation); unit: millivolt (mV)
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 166 | 170
millivolt (mV) | 3.0 (1.3) | 3.1 (1.4)

16. Secondary Outcome: Ventricular Sensed Amplitude
Description: Average ventricular sensed amplitude.
Time Frame: 3 or 4 months post-implant
Measure: Mean (Standard Deviation); unit: millivolt (mV)
Groups:
- 5086 MRI Lead: The MRI group underwent a one-hour MRI scan at 9-12 weeks post-implant.
Arm/Group | 5086 MRI Lead | Control Group
Number analyzed (Participants) | 179 | 176
millivolt (mV) | 10.1 (5.0) | 10.2 (5.2)

ADVERSE EVENTS:
Time Frame: Up to 31 months.
Description: Serious AE:
  AE that led to death, or led to worse health that resulted in: life-threatening illness or injury; a permanent impairment of a body function; hosp.; medical or surgery to prevent permanent impairment to body structure or a body function.
  2 more MRI and 1 more control participants here due to a later freeze of adverse event data.
Groups:
- Non-randomized: Some subjects were enrolled, but either did not receive a system, or received only a partial system, and were not randomized. Their adverse events were collected until they exited the study.
Arm/Group | MRI Group | Control Group | Non-randomized
Serious Adverse Events (participants affected / at risk) | 117/260 | 77/207 | 3/20
Other Adverse Events (participants affected / at risk) | 24/260 | 19/207 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI Group (N=260) | Control Group (N=207) | Non-randomized (N=20)
Atrial fibrillation (Cardiac disorders) | 13 (17) | 5 (5) | 1 (1)
Lead dislodgement (Injury, poisoning and procedural complications) | 12 (12) | 6 (6) | 0 (0)
Chest pain (General disorders) | 8 (8) | 7 (7) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 5 (5) | 2 (2)
Elevated pacing threshold (Injury, poisoning and procedural complications) | 6 (6) | 2 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 6 (7) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 5 (5) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 7 (7) | 0 (0) | 0 (0)
Plural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Failure to capture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (2) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Pulmoary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (2) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cardiac perforation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Implant site haematoma (General disorders) | 0 (0) | 2 (2) | 0 (0)
Knee arthoplasty (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess soft tissue (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerotic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker revision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecytitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholinergic syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cytocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Endometrial disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocoocal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fibroadenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gliobastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Implant site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inappropriate device stimulation of tissue (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Medical device complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pacemaker generated arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI Group (N=260) | Control Group (N=207) | Non-randomized (N=20)
Atrial fibrillation (Cardiac disorders) | 24 (27) | 19 (24) | 0 (0)

LIMITATIONS AND CAVEATS:
Comparisons with a historical control (5076 Lead) were performed for secondary objectives #11-#16, however the results database is currently only designed to allow for reporting of participants specifically enrolled as part of this protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No